CLINICAL TRIAL: NCT04863508
Title: Application of the HeartGuide Blood Pressure Watch Monitor to Identify Masked Uncontrolled Hypertension in Hypertensive Patients With Different Cardiovascular Risks In Taiwan.
Brief Title: Wearable Blood Pressure Devices to Identify Masked Uncontrolled Hypertension.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Other Study IDs: 109-029-E
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hypertension,Essential; Hypertension, Masked
Keywords: home blood pressure monitoring; wearable blood pressure device; masked uncontrolled hypertension
MeSH Terms: conditions — Essential Hypertension; Masked Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low-risk hypertensive patients: Patients without diabetes, chronic kidney disease, hypertension-mediated organ damage, or established cardiovascular diseases
- With-risk hypertensive patients: Patients with diabetes, chronic kidney disease, hypertension-mediated organ damage, but without established cardiovascular diseases
- Hypertensive patients with cardiovascular diseases: Patients with established cardiovascular diseases

SUMMARY:
Uncontrolled out-of-office blood pressure (BP), measured by either home BP monitoring (HBPM) or ambulatory BP monitoring, has been shown to predict higher cardiovascular risk. However, HBPM could not identify daytime BP surge, which leads to underestimation of future risk among treated hypertensive individuals.

HeartGuide provides validated out-of-office BP measurements, along with activity/sleep recordings. The present study is designed to examine whether BP monitoring with the HeartGuide could identify masked uncontrolled hypertension in controlled hypertensive patients based on office BP. We will enroll hypertensive patients with controlled office BP according to their cardiovascular risk profile. We will also examine prevalence of post-prandial BP changes and BP variability using HeartGuide.

DETAILED DESCRIPTION:
Recent hypertension guidelines stressed the importance of out-of-office BP monitoring. Ambulatory BP (ABPM) and home BP monitoring (HBPM) both predict future cardiovascular events better than office BP. Masked hypertension is an important issue. As revealed by recent studies, daytime BP surge can result in greater target organ damage for high-risk hypertensive individuals.

Previous trials such as TASMINH2 and TASMINH-SR study showed positive effects of HBPM on BP control in hypertensive patients. However, several issues preclude perfect applications of HBPM. For example, HBPM could not provide BP recordings during activity or at night-time. In addition, the currently recommended time schedule for HBPM may be insufficient for detecting daytime surge especially among high-risk individuals. Wearable BP devices seem to fill in this gap as a novel approach of out-of-office monitoring.

HeartGuide, the new watch BP monitor, was recently validated to provide accurate BP measurements. It could provide incremental knowledge with potentially larger numbers of recordings. The primary objective of this study is to unveil uncontrolled masked hypertension with HeartGuide, particularly for those undetected with current office BP and HBPM. A second objective is to assess diurnal BP trends and BP variability.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign informed consent form
* Currently taking anti-hypertensive therapy for more than 3 months
* Drugs are unchanged during the study period
* Office BP below 140/90 mmHg at least one visit

Exclusion Criteria:

* Diagnosed with terminal illness
* End-stage renal disease requiring lifelong dialysis treatment
* Patients with impaired performance status (ECOG >= 2)
* Women undergoing or expecting pregnancy during the study period
* Resistant hypertension (taking more than 4 kinds of anti-hypertensive drugs)
* Known atrial or ventricular arrhythmia
* Wrist circumference out-of range between 13.5 to 21.5 cm

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants routinely treated at out-patient clinics for hypertension are to be enrolled after informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of masked uncontrolled hypertension | during 3-month follow-up period
  measured BP>=135/85 mmHg by wearable BP devices or average BP>=130/80 mmHg by ambulatory BP monitor

OTHER OUTCOMES:
Newly diagnosed left ventricular hypertrophy by echocardiography | at 3-month follow-up
  left ventricular mass index>=115 g/m2(men) or >=95 g/m2(women)
Occurrence of post-prandial BP change | during 3-month follow-up period
  measured BP drop >= 20 mmHg pre- and post-meal
BP variability | during 3-month follow-up period
  coefficient of variation of all measured BP values by either HeartGuide or ambulatory BP monitor

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoshide S, Cheng HM, Huang Q, Park S, Park CG, Chen CH, Wang JG, Kario K; Characteristics On the ManagEment of Hypertension in Asia - Morning Hypertension Discussion Group (COME Asia MHDG). Role of ambulatory blood pressure monitoring for the management of hypertension in Asian populations. J Clin Hypertens (Greenwich). 2017 Dec;19(12):1240-1245. doi: 10.1111/jch.13086. Epub 2017 Aug 22. PMID 28834205
- [Background] McManus RJ, Mant J, Bray EP, Holder R, Jones MI, Greenfield S, Kaambwa B, Banting M, Bryan S, Little P, Williams B, Hobbs FD. Telemonitoring and self-management in the control of hypertension (TASMINH2): a randomised controlled trial. Lancet. 2010 Jul 17;376(9736):163-72. doi: 10.1016/S0140-6736(10)60964-6. Epub 2010 Jul 8. PMID 20619448
- [Background] McManus RJ, Mant J, Haque MS, Bray EP, Bryan S, Greenfield SM, Jones MI, Jowett S, Little P, Penaloza C, Schwartz C, Shackleford H, Shovelton C, Varghese J, Williams B, Hobbs FD, Gooding T, Morrey I, Fisher C, Buckley D. Effect of self-monitoring and medication self-titration on systolic blood pressure in hypertensive patients at high risk of cardiovascular disease: the TASMIN-SR randomized clinical trial. JAMA. 2014 Aug 27;312(8):799-808. doi: 10.1001/jama.2014.10057. PMID 25157723
- [Background] Kuwabara M, Harada K, Hishiki Y, Kario K. Validation of a wrist-type home nocturnal blood pressure monitor in the sitting and supine position according to the ANSI/AAMI/ISO81060-2:2013 guidelines: Omron HEM-9600T. J Clin Hypertens (Greenwich). 2019 Apr;21(4):463-469. doi: 10.1111/jch.13464. Epub 2019 Jan 4. PMID 30609129